CLINICAL TRIAL: NCT00963131
Title: High-dose Antioxidants for Central Serous Chorioretinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Associated professor Mansing Ratanasukon, MD, Department of Ophthalmology, Faculty of medicine, Prince of Songkla university
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC 47/362-023; PSU 2547 (Other: Prince of Songkla University)
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-12

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Central serous chorioretinopathy,antioxidants
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antioxidant tablets (Experimental): the study arm received antioxidant tablets (Icaps) for 3 months or until the resolution of the disease
  Interventions: Drug: antioxidants tablets
- placebo tablets (Placebo Comparator): the control arm received placebo tablets for 3 months or until the resolution of the disease
  Interventions: Drug: antioxidants tablets

INTERVENTIONS:
Drug: antioxidants tablets — vitamin A 6600 IU, vitamin C 400 mg, vitamin E 150 IU, riboflavin 10 mg, zinc 60 mg, copper 4 mg, selenium 40 mg, manganese 4 mg and lutein/zeaxanthin 4000 micrograms.
  Other Names: Icaps

SUMMARY:
Central serous chorioretinopathy (CSC) is the serous neurosensory detachment that usually involves the macular area. It is common in patients between 30-50 years old and effects male more often than female with the ratio of 5-10. The common risk factors are psychologic stress, type A personality, systemic steroid use, hypertension and pregnancy. The treatment is usually observation especially in the first three-months. The laser or photodynamic therapy should be considered when the condition does not improve after that time. Nevertheless, the pathogenesis of CSC is still not well understood but the study from indocyanine green angiography showed the choroidal vascular hyperpermeability and abnormal leakage. The causes of this abnormality are supposed to be from nitric oxide, prostaglandins or even free oxidative radicals. From this hypothesis, the oxidative process might be involved in the pathogenesis of the disease especially in the early stage. This study is to determine the effect of antioxidants drugs in the acute stage of CSC and to determine whether they can improve the outcomes of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. patients with acute central serous chorioretinopathy within 6 weeks of onset
2. age between 30-50 years
3. new or recurrent attack (the symptom-free period should longer than 6 months)
4. fluorescein angiography (FA) confirmed the diagnosis with the inkblot or smoke-stack leakage and the optical coherence tomography (OCT) showed definite subretinal fluid
5. patients' ability for proper follow up.

Exclusion Criteria:

1. chronic central serous chorioretinopathy(longer than 6 weeks)
2. complicated central serous chorioretinopathy such as secondary choroidal neovascularization (CNV) that detected from FA
3. pregnancy, steroid user and patients that contraindicated for high dose antioxidants therapy such as heavy smokers, lung cancer, thyrotoxicosis, renal stone and anemia (hematocrit less than 30%).

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-12; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
visual acuity and central macular thickness | 6 months

SECONDARY OUTCOMES:
fluorescein leakage at the third month | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mansing - Ratnasukon, MD, Principal Investigator — Department of Ophthalmology, Faculty of medicine, Prince of Songkla university, Hat yai, Songkhla province, Thailand 90110
Locations (1):
- Department of Ophthalmology, Faculty of medicine, Prince of Songkla university, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203